CLINICAL TRIAL: NCT05056155
Title: Systane Complete Multi-symptom Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEC262-P002
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Dry Eye Disease
Keywords: Eye drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systane Complete (Experimental): First dose of Systane Complete in both eyes on Day 0, followed by Systane Complete self-administered 4 times daily for 28 days
  Interventions: Other: Systane Complete

INTERVENTIONS:
Other: Systane Complete — Propylene glycol 0.6% eye drops for replenishing deficiencies in both the lipid and aqueous layers of the tear film
  Other Names: Systane® Complete Lubricant Eye Drops

SUMMARY:
The purpose of this study is to demonstrate effective symptom relief with the use of Systane Complete among subjects with dry eye disease (DED).

DETAILED DESCRIPTION:
Subjects will be expected to attend a screening/baseline visit and one additional visit at Day 28 (± 2 days), with a telephone call visit conducted at Day 14 (± 2 days). Individual duration of subject participation will be approximately 28 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form.
* Willing and able to attend all study visits as required per protocol.
* Have dry eye symptoms as specified in the protocol.
* Willing to discontinue use of all habitual artificial tear supplements for the entire study duration.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Ocular conditions as specified in the protocol.
* Contact lens use within one week prior to screening visit.
* Use of medications as specified in the protocol.
* Pregnant or breast feeding.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Change from Baseline at Day 28 in IDEEL-SB Question "Sore" | Baseline (Day 0), Day 28
  The Impact of Dry Eye on Everyday Life - Symptoms Bother (IDEEL-SB) is a patient-reported outcome measures questionnaire designed to assess symptoms of dry eye disease. Subjects will respond to the question, "OVER THE LAST TWO WEEKS, how much did the following symptom bother you: Sore Eyes?" using a 0-4 Likert-type scale, where 0 = "I did not have this symptom/Not applicable" and 4 = Very Much. A negative change value will represent perceived improvement.
Change from Baseline at Day 28 in IDEEL-SB Question "Stinging" | Baseline (Day 0), Day 28
  Subjects will respond to the question, "OVER THE LAST TWO WEEKS, how much did the following symptom bother you: Stinging Eyes?" using a 0-4 Likert-type scale, where 0 = "I did not have this symptom/Not applicable" and 4 = Very Much. A negative change value will represent perceived improvement.
Change from Baseline at Day 28 in IDEEL-SB Question "Burning" | Baseline (Day 0), Day 28
  Subjects will respond to the question, "OVER THE LAST TWO WEEKS, how much did the following symptom bother you: Burning Eyes?" using a 0-4 Likert-type scale, where 0 = "I did not have this symptom/Not applicable" and 4 = Very Much. A negative change value will represent perceived improvement.
Change from Baseline at Day 28 in IDEEL-SB Question "Tired Eyes" | Baseline (Day 0), Day 28
  Subjects will respond to the question, "OVER THE LAST TWO WEEKS, how much did the following symptom bother you: Tired Eyes?" using a 0-4 Likert-type scale, where 0 = "I did not have this symptom/Not applicable" and 4 = Very Much. A negative change value will represent perceived improvement.
Change from Baseline at Day 28 in DEQ-5 Question "Watery" | Baseline (Day 0), Day 28
  The Dry Eye Questionnaire-5 (DEQ-5) is a patient-reported outcome measures questionnaire designed to assess symptoms of dry eye disease. Subjects will respond to the question, "During a typical day in the past month, how often did your eyes look or feel excessively watery?" using a 0-4 Likert-type scale, where 0 = Never and 4 = Constantly. A negative change value will represent perceived improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Ocular Health, Study Director — Alcon Research, LLC
Locations (4):
- United States (4):
  - Alcon Investigator 1455, Kansas City, Missouri
  - Alcon Investigator 8046, Granville, Ohio
  - Alcon Investigator 6313, Powell, Ohio
  - Alcon Investigator 8175, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bickle K, Miller JR, Tauber J, Awisi-Gyau D. Multi-symptom Relief with Propylene Glycol-Hydroxypropyl-Guar Nanoemulsion Lubricant Eye Drops in Subjects with Dry Eye Disease: A Post-Marketing Prospective Study. Ophthalmol Ther. 2024 Feb;13(2):481-494. doi: 10.1007/s40123-023-00853-3. Epub 2023 Dec 11. PMID 38079084